CLINICAL TRIAL: NCT05448456
Title: Use of Tranexamic Acid After Vaginal Delivery with Episiotomy a RCT Placebo Control Trail
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Principal Investigator, Eran Brazilay, MD PhD, Head of the obstetric and gynecologic ultrasound unit, Assuta Ashdod Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0138-21-AA
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-09

CONDITIONS: Episiotomy Wound; Anemia; Early Postpartum Hemorrhage; Hemoglobin
MeSH Terms: conditions — Anemia; Postpartum Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hexakakapron group (Active Comparator): women with an episiotomy after vaginal delivery
  Interventions: Drug: Tranexamic acid
- control group (Placebo Comparator): women with an episiotomy after vaginal delivery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — 1 gram of tranexamic acid in 100 ml of 0.9% normal saline
  Other Names: Hexakapron
  Arms: Hexakakapron group
Drug: Placebo — 100 ml of 0.9% normal saline
  Other Names: saline
  Arms: control group

SUMMARY:
The objective of this study is to assess the effect of TA treatment on decline in Hb levels following vaginal delivery with an episiotomy, compared to a control group not receiving TA.

DETAILED DESCRIPTION:
Vaginal delivery is often characterized by excessive blood loss. Normal range of blood loss in uncomplicated vaginal delivery is up to 500 ml. Despite this, most women can adapt due to hemodynamic changes that occur during pregnancy Several factors during labor can promote major blood loss that may be defined as post-partum hemorrhage (PPH) Early PPH (E-PPH) is defined by the World Health Organization as "blood loss from the birth canal in excess of 500 ml during the first 24 hours after delivery E-PPH occurs in up to 6% of births and it is one of the main causes of maternal morbidity and mortality accounting for about 25% of maternal deaths worldwide Among morbidities, E-PPH can lead to post-partum anemia (PPA). PPA incidence is estimated between 50%-80% of women PPA is defined as level of hemoglobin (Hb) of 11 gr/dl one week after delivery Anemia is associated with fatigue, post-partum depression and is a significant health problem in women during the reproductive age .

One of the major causes of E-PPH is perineal trauma. Perineal trauma is present in up to 85% of births either due to an episiotomy or spontaneous tear or a combination of them both During the the second stage of labor, the midwife or the obstetrician may need to make a surgical incision (episiotomy) to increase the diameter of the vaginal outlet and facilitate the baby's birth This procedure is done with scissors or scalpel and requires repair by suturing (14). In the United States, episiotomy rate was 11.6% in 2012 In a study published by Alvarez et al in 2017, the average reduction in Hb was 1.46 ± 1.09 g/dl following vaginal delivery with a second degree tear but without an episiotomy and 2.07 ± 1.24 following vaginal delivery with an episiotomy and no perineal tear. The greatest reduction in Hb occurred among women with episiotomy and a third or fourth degree tear with a decrease of 3.1 ± 1.32 g/dl.

Different strategies have been described for preventing and treatment PPH, including active management of the third stage of labor, among them uterine massage and controlled cord traction in addition to oxytocin and the use of Tranexamic acid (TA) as PPH treatment Tranexamic acid (TA) is a lysine analog, which acts as an antifibrinolytic via competitive inhibition to the binding of plasmin and plasminogen to fibrin. TA reaches peak plasma concentration immediately after intravenous administration A meta-analysis evaluated the use of tranexamic acid after vaginal delivery for prevention of primary PPH. When used as prophylaxis within 10 min after vaginal delivery usually at the dose of 1 g IV, in addition to standard prophylaxis with oxytocin, tranexamic acid reduced the risk of primary PPH and the mean post-partum blood loss However there are no studies that evaluated the impact of TA on blood loss after vaginal deliveries with an episiotomy.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18-45
2. 37-42 weeks gestation
3. Singleton pregnancy
4. Cephalic presentation

Exclusion Criteria:

1. Any contra-indication for vaginal birth
2. PPH risk factors

   1. Dysfunctional labor
   2. Over distended uterus (macrosomia ,Polyhydramnios,multiple gestation)
   3. Grand multiparity
   4. Chorioamnionitis
   5. Precipitous labor
   6. Operative delivery
   7. Prolonged second stage
3. Previous pph
4. Preeclampsia
5. Placental abruption
6. Previous cesarean delivery
7. Thrombophilia or coagulopathy
8. Allergy to TA

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Delta Hb levels | 24 hours from delivery
  Delta-Hb (Hb level prior delivery - Hb levels 24 h after birth)

SECONDARY OUTCOMES:
PPH rate | 24 hours from delivery
  early post partum hemorrhage
Uterotonics use | 24 hours from delivery
  Use of additional uterotonics drugs(other than oxytocin)- dichotomies scale, yes or no
Blood transfusion | 72 hours from delivery
  Use of Blood packed cells during hospitalization, dichotomies scale - yes or no
hospital admission | 120 hours from delivery
  Number of hospital admission days

CONTACTS AND LOCATIONS:
Overall Officials: Atara De Porto Amrany, MD, Principal Investigator — Samson Assuta Ashdod University Hospital
Locations (1):
- Assuta ashdod, Ashdod, Shfela, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carbillon L, Uzan M, Uzan S. Pregnancy, vascular tone, and maternal hemodynamics: a crucial adaptation. Obstet Gynecol Surv. 2000 Sep;55(9):574-81. doi: 10.1097/00006254-200009000-00023. PMID 10975484
- [Background] Kramer MS, Berg C, Abenhaim H, Dahhou M, Rouleau J, Mehrabadi A, Joseph KS. Incidence, risk factors, and temporal trends in severe postpartum hemorrhage. Am J Obstet Gynecol. 2013 Nov;209(5):449.e1-7. doi: 10.1016/j.ajog.2013.07.007. Epub 2013 Jul 16. PMID 23871950
- [Background] Rossen J, Okland I, Nilsen OB, Eggebo TM. Is there an increase of postpartum hemorrhage, and is severe hemorrhage associated with more frequent use of obstetric interventions? Acta Obstet Gynecol Scand. 2010 Oct;89(10):1248-55. doi: 10.3109/00016349.2010.514324. PMID 20809871
- [Background] Sosa CG, Althabe F, Belizan JM, Buekens P. Risk factors for postpartum hemorrhage in vaginal deliveries in a Latin-American population. Obstet Gynecol. 2009 Jun;113(6):1313-1319. doi: 10.1097/AOG.0b013e3181a66b05. PMID 19461428